CLINICAL TRIAL: NCT00771095
Title: Pounds Off Digitally Study: A Podcasting Weight Loss Intervention
Acronym: POD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: UNC Lineberger's Cancer Control Education Program (Unknown)
Responsible Party: Gabrielle Turner-McGrievy, UNC-Chapel Hill
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0430-03
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Weight Loss
Keywords: weight loss; elaboration; self efficacy
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (available) podcast (Active Comparator)
  Interventions: Behavioral: podcasting
- Enhanced podcast (Experimental)
  Interventions: Behavioral: podcasting

INTERVENTIONS:
Behavioral: podcasting

SUMMARY:
Participants in both the existing and enhanced podcast groups will lose weight. The enhanced podcasting group will have a greater increase in weight loss, elaboration, self-efficacy, and perceived control than the existing podcast group.

DETAILED DESCRIPTION:
We will conduct a weight loss intervention study among adults. Using the weight loss podcast that receives the highest rating from a previous content analysis, we will conduct an intervention comparing the best existing weight loss podcast to an enhanced podcast. The enhanced podcast will be based on theoretical constructs that have been shown to be effective in producing weight loss in other research studies. We will then evaluate the effectiveness of podcasting to promote weight loss in adults. Weight change from baseline to 12-weeks and changes in psychosocial measures will be used to assess differences between the existing podcast, enhanced podcast, and control conditions. In conclusion, this research study aims to find innovative and inexpensive ways to help people lose weight. Podcasting has the possibility of reaching a wide range of age and ethnic groups and will allow people to receive weight loss information when and where it is convenient for them.

ELIGIBILITY:
Inclusion Criteria:

be 18-50 years old be overweight or obese (BMI between 25-35) but not severely or morbidly obese live in the Chapel Hill area be able to attend an introduction meeting and weigh-in before the study and a weigh-in after the study have access to the Internet and a computer with a sound card have a working MP3 player that can connect to a computer have access to a scale be willing to be randomized to any group

Exclusion Criteria:

smoker current major health or psychiatric diseases, drug or alcohol dependency, uncontrolled thyroid conditions, eating disorder, or pregnancy participation in a weight loss program or taking weight loss medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
weight | 12 weeks

SECONDARY OUTCOMES:
elaboration | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Turner-McGrievy GM, Campbell MK, Tate DF, Truesdale KP, Bowling JM, Crosby L. Pounds Off Digitally study: a randomized podcasting weight-loss intervention. Am J Prev Med. 2009 Oct;37(4):263-9. doi: 10.1016/j.amepre.2009.06.010. PMID 19765496